CLINICAL TRIAL: NCT03251092
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PTI-808 in Healthy Adult Subjects and in Adults With Cystic Fibrosis
Brief Title: Study Designed to Assess the Safety, Tolerability and PK of PTI-808 in Healthy Volunteers and in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PTI-808-01
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteer - Complete; Cystic Fibrosis - Complete

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- SAD PTI-808 Active (Active Comparator): Three cohorts of SAD are planned for evaluation where subjects will be randomized to PTI-808 or placebo.
  Interventions: Drug: PTI-808
- SAD PTI-808 Placebo (Placebo Comparator): Three cohorts of SAD are planned for evaluation where subjects will be randomized to PTI-808 or placebo.
  Interventions: Drug: Placebo
- MAD PTI-808 Active (Active Comparator): Three cohorts of MAD are planned for evaluation where subjects will be randomized to PTI-808 or placebo.
  Interventions: Drug: PTI-808
- MAD PTI-808 Placebo (Placebo Comparator): Three cohorts of MAD are planned for evaluation where subjects will be randomized to PTI-808 or placebo.
  Interventions: Drug: Placebo
- FE PTI-808 Active (Active Comparator): Subjects will be randomized to Fed or Fasted on Days 1 and 12. Follow up visits will occur 7 days post Day 12 dose.
  Interventions: Drug: PTI-808
- FE PTI-808 Placebo (Placebo Comparator): Subjects will be randomized to Fed or Fasted on Days 1 and 12. Follow up visits will occur 7 days post Day 12 dose.
  Interventions: Drug: Placebo
- Part 2 PTI-808 + PTI-801 + PTI-428 Active (Experimental): One cohort is planned where subjects will be randomized to either the triple active arm (dosed with PTI 808+PTI 801+PTI 428) OR placebo arm.
  Interventions: Drug: PTI-808; Drug: PTI-428; Drug: PTI-801
- Part 2 matching Placebos (Placebo Comparator): In all three cohorts in part 2, subjects will be randomized to active drug or placebo. The placebo arm for all cohorts consists of placebo capsules matching PTI-808+PTI-801+PTI-428.
  Interventions: Drug: Placebo
- Part 2 dual active arm PTI-801+PTI-428+ PTI-808 placebo (Experimental): One cohort is planned where subjects are randomized to either 808 placebo + dual active arm (dosed with placebo matching PTI 808 plus PTI 801 + PTI 428) OR placebo arm.
  Interventions: Drug: Placebo; Drug: PTI-428; Drug: PTI-801
- Part 2 dual active arm PTI-801+PTI-808+PTI-428 placebo (Active Comparator): One cohort is planned where subjects are randomized to either 428 placebo + dual active arm (dosed with placebo matching PTI 428 plus PTI 808 and PTI 801) OR placebo arm.
  Interventions: Drug: PTI-808; Drug: Placebo; Drug: PTI-801
- Part 3 CF MAD PTI-808 + PTI-801 + PTI-428 (Active Comparator): In all cohorts in Part 3, subjects will be will be randomized to receive 7 days of PTI-808 or placebo followed by 14 days of co-administration of PTI-808+PTI-801+PTI-428 or matching placebos. A follow-up will occur on Day 28.
  Interventions: Drug: PTI-808; Drug: PTI-428; Drug: PTI-801
- Part 3 CF MAD PTI-808 placebo+PTI-801 placebo+PTI-428 placebo (Placebo Comparator): In all cohorts in Part 3, subjects will be randomized to receive 7 days of PTI-808 or placebo followed by 14 days of co-administration of PTI-808+PTI-801+PTI-428 or matching placebos. A follow-up will occur on Day 28.
  Interventions: Drug: Placebo
- Part 4 CF PTI-808 + PTI-801 + PTI-428 (Active Comparator): In cohorts 3 & 4 subjects will be randomized to receive PTI-808 + PTI-801 with or without PTI-428 or matching placebos. A follow-up will occur on Day 42.
  Interventions: Drug: PTI-808; Drug: PTI-428; Drug: PTI-801
- Part 4 CF PTI-808 + PTI-801 + PTI-428 placebo (Active Comparator): In cohorts 3 & 4, subjects will be randomized to receive PTI-808 + PTI-801 with or without PTI-428 or matching placebos. A follow-up will occur on Day 42.
  Interventions: Drug: PTI-808; Drug: PTI-801
- Part 4 CF PTI-808 placebo + PTI-801 placebo + PTI-428 placebo (Placebo Comparator): In cohorts 3 & 4, subjects will be randomized to receive PTI-808 + PTI-801 with or without PTI-428 or matching placebos. A follow-up will occur on Day 42.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTI-808 — Active
  Arms: FE PTI-808 Active; MAD PTI-808 Active; Part 2 PTI-808 + PTI-801 + PTI-428 Active; Part 2 dual active arm PTI-801+PTI-808+PTI-428 placebo; Part 3 CF MAD PTI-808 + PTI-801 + PTI-428; Part 4 CF PTI-808 + PTI-801 + PTI-428; Part 4 CF PTI-808 + PTI-801 + PTI-428 placebo; SAD PTI-808 Active
Drug: Placebo — Placebo
  Arms: FE PTI-808 Placebo; MAD PTI-808 Placebo; Part 2 dual active arm PTI-801+PTI-428+ PTI-808 placebo; Part 2 dual active arm PTI-801+PTI-808+PTI-428 placebo; Part 2 matching Placebos; Part 3 CF MAD PTI-808 placebo+PTI-801 placebo+PTI-428 placebo; Part 4 CF PTI-808 placebo + PTI-801 placebo + PTI-428 placebo; SAD PTI-808 Placebo
Drug: PTI-428 — Active
  Arms: Part 2 PTI-808 + PTI-801 + PTI-428 Active; Part 2 dual active arm PTI-801+PTI-428+ PTI-808 placebo; Part 3 CF MAD PTI-808 + PTI-801 + PTI-428; Part 4 CF PTI-808 + PTI-801 + PTI-428
Drug: PTI-801 — Active
  Arms: Part 2 PTI-808 + PTI-801 + PTI-428 Active; Part 2 dual active arm PTI-801+PTI-428+ PTI-808 placebo; Part 2 dual active arm PTI-801+PTI-808+PTI-428 placebo; Part 3 CF MAD PTI-808 + PTI-801 + PTI-428; Part 4 CF PTI-808 + PTI-801 + PTI-428; Part 4 CF PTI-808 + PTI-801 + PTI-428 placebo

SUMMARY:
Part 1 of this trial will enroll healthy volunteers into a single ascending dose (SAD), multiple ascending dose (MAD), and Food Effect (FE) treatment groups.

The SAD treatment group is comprised of at least 3 ascending dose level cohorts where healthy adult subjects will be randomized to receive a single dose of either PTI-808 or placebo and will be followed for 7 days post dose. A safety review committee (SRC) will convene after the completion of each cohort to evaluate safety and pharmacokinetic (PK) data.

Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 ascending dose level cohorts where subjects will be randomized to receive either PTI-808 or placebo daily for 7 days and will be followed for 7 days after receiving the last dose.

Also following the conclusion of the respective SAD level dose groups, healthy adult subjects will participate in the FE treatment group.

Part 2 of this will enroll healthy volunteers to assess the safety, tolerability, and PK of PTI 808 co administered with PTI 801 and PTI 428 to HVs with daily dosing for 7 consecutive days.

Part 3 will enroll adult subjects with cystic fibrosis (CF) into a MAD treatment group consisting of 2 cohorts. Subjects will receive PTI-808 co-administered with PTI-801 and PTI-428. PTI-808 will be administered daily for 7 consecutive days followed by PTI-808 + PTI-801 + PTI-428 administered daily for 14 consecutive days.

Part 4 will enroll adult subjects with cystic fibrosis (CF) into 28-day cohorts. Subjects will receive PTI-808 co-administered with PTI-801 with or without PTI-428 versus matching placebo.

DETAILED DESCRIPTION:
Part 1 of this trial will enroll healthy volunteers into a single ascending dose (SAD), multiple ascending dose (MAD), and Food Effect (FE) treatment groups.

The SAD treatment group is comprised of at least 3 ascending dose level cohorts where healthy adult subjects will be randomized to receive a single dose of either PTI-808 or placebo and will be followed for 7 days post dose.

The MAD treatment group is comprised of 3 ascending dose level cohorts where subjects will be randomized to receive either PTI-808 or placebo daily for 7 days and will be followed for 7 days after receiving the last dose.

Following the conclusion of the respective SAD level dose groups the food effect portion of the study will be initiated and subjects will be randomized to receive an initial single dose of PTI-808 either after an overnight fast of at least 10 hours (fasted group) or after an overnight fast of at least 10 hours followed the consumption of a high fat high calorie meal (fed group). After a 10 day washout period, subjects will cross over to the opposite group and receive a second dose of PTI-808. Subjects will be followed for up to 7 days following dosing.

Part 2 of this will enroll healthy volunteers to assess the safety, tolerability, and PK of PTI 808 co administered with PTI 801 and PTI 428 to HVs with daily dosing for 7 consecutive days.

Part 3 - Part 3 will enroll adult subjects with CF to assess the safety, tolerability, and PK of multiple ascending doses of PTI-808 co-administered with PTI-801 and PTI-428. Subjects will receive 7 days of PTI-808 or placebo followed by 14 days of PTI-808 or placebo co-administered with PTI-801+PTI-428 or matching placebos.

Part 4 - Part 4 will assess the safety, tolerability, PK, and the effects of PTI-808 co-administered with PTI-801 with or without PTI-428 over a 28-day treatment period in CF subjects who are either homozygous for the F508del CFTR genotype or are heterozygous for the F508del CFTR genotype. Subjects will be randomized to receive treatment with PTI-808 co-administered with PTI-801 with or without PTI-428 versus matching placebo.

ELIGIBILITY:
Part 1 and Part 2 Inclusion Criteria:

1. Adults aged 18 to 55 years old, inclusive, at the time of informed consent
2. Body mass index ≥18 and <30 kg/m2
3. Subject must be a non-smoker and non-tobacco user for a minimum of 30 days prior to screening and for the duration of the study.
4. Subject understands the full nature and purpose of the study, including possible risks and side effects, and is willing and able to comply with all compulsory study procedures and provides informed consent/permission prior to any study procedures being performed.
5. Females of childbearing potential and males capable of fathering a child must meet the contraception requirements

Part 1 & Part 2 Exclusion Criteria:

1. History or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the investigator
2. Prolonged QT interval with Fridericia's correction >450 msec at screening
3. Abnormal liver function as defined by aspartate transaminase (AST), alanine transaminase (ALT), or bilirubin >1.5× the upper limit of the normal range
4. Abnormal renal function at screening defined as creatinine clearance <90 mL/min using the Cockroft-Gault equation
5. Clinically significant screening results that would exclude subject from the study (e.g., medical histories, PE, ECGs, vital signs, and laboratory profiles) as deemed by the investigator
6. Participation in another clinical study or treatment with an investigational agent within 30 days or five half-lives, whichever is longer, prior to Study Day 1
7. History of cancer within the past 5 years (excluding non-melanoma skin cancer)
8. History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
9. Positive urine screen for prohibited drugs (cocaine, cannabinoids, nicotine [urine cotinine is the detection mechanism for nicotine], opiates, barbiturates, amphetamines, and benzodiazepines) or positive alcohol test at screening
10. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb)
11. Clinically significant infection within 3 months of screening as determined by the investigator
12. Known or suspected hypersensitivity or idiosyncratic reaction to study medication or any components thereof
13. Has donated blood within 3 months of screening or plans to donate blood within 3 months of study completion
14. Pregnant or nursing women
15. Any conditions that, in the opinion of the investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study
16. Use of prohibited medications within 14 days prior to dosing of study drug

Part 3 CF Inclusion Criteria:

1. Confirmed diagnosis of CF with the F508del/F508del genotype
2. Forced expiratory volume in 1 second (FEV1) 40-90% predicted, inclusive
3. Non-smoker and non-tobacco user for a minimum of 30 days prior to screening

Part 3 CF Exclusion Criteria:

1. Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Study Day 1
2. History of cancer within the past 5 years (excluding cervical cancer in situ with curative therapy for at least one year prior to screening and non-melanoma skin cancer)
3. History of organ transplantation
4. Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (as determined by the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 14 days of Day 1
5. Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®)) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to Day 1
6. History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
7. Pregnant or nursing women
8. Currently taking or has taken a CFTR modulator within 30 days prior to initial dose of study drugs

Part 4 CF Inclusion Criteria:

1. Confirmed diagnosis of CF with either the F508del CFTR homozygous genotype on record or for heterozygote subjects, only one copy of the F508del CFTR mutation on record
2. Forced expiratory volume in 1 second (FEV1) 40-90% predicted, inclusive
3. Non-smoker and non-tobacco user for a minimum of 30 days prior to screening

Part 4 CF Exclusion Criteria:

1. Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Study Day 1
2. History of cancer within the past 5 years (excluding cervical cancer in situ with curative therapy for at least one year prior to screening and non-melanoma skin cancer)
3. History of organ transplantation
4. Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (as determined by the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 28 days of Day 1
5. Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®)) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days of Day 1
6. History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
7. Pregnant or nursing women
8. Currently taking or has taken a CFTR modulator within 14 days prior to the screening visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Part 1 SAD and MAD: Adverse Events | Baseline to up to 14 days
  Safety and tolerability measure by number of subjects who experience adverse events
Part 1 SAD and MAD: Physical Exams | Baseline to up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in physical examinations
Part 1 SAD and MAD: The number of subjects who experience potential clinically significant changes in vital signs | Baseline to up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in vital signs
Part 1 SAD and MAD: ECGs | Baseline to up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in ECGs
Part 1 SAD and MAD: The number of subjects who experience potential clinically significant changes in safety labs | Baseline to up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in safety labs
Part 1 SAD and FE: terminal half life | Through 72 hours post dose
  Apparent terminal half-life (t1/2) of single oral dose
Part 1 SAD and FE : Tmax | Through 72 hours post dose
  Time to reach maximum plasma concentration (Tmax) of single oral dose
Part 1 SAD and FE: Cmax | Through 72 hours post dose
  Maximum plasma concentration (Cmax) of single oral dose
Part 1 SAD : AUC | Through 24 hours post dose
  Area under the concentration-time curve from time 0 to 24 hours post dose (AUC 0-24) of single oral dose
Part 1 SAD and FE: AUC0 | Through 72 hours post dose
  AUC from time 0 to time of last measurable concentration (AUC0-last) of single oral dose
Part 1 SAD and FE: AUC0-inf | Through 72 hours post dose
  AUC from time 0 to infinity (AUC0-inf) of single dose
Part 1 MAD: t1/2 | Through 72 hours post dose
  t1/2 of multiple oral dose
Part 1 MAD: Tmax | Through 72 hours post dose
  Tmax of multiple oral doses
Part 1 MAD: Cmax | Through 72 hours post last dose
  Cmax of multiple oral doses
Part 1 MAD: AUC0-24 | Through 24 hours post last dose
  AUC0-24 of multiple oral dose
Part 1 MAD: AUC0-last | Through 72 hours post last dose
  AUC0-last of multiple oral doses
Part 1 MAD: Urine | Through 24 hours post last dose
  Cumulative amount of PTI-808 excreted unchanged in urine (Ae) as appropriate of multiple oral doses
Part 1 MAD: CLR | Through 24 hours post dose
  Renal clearance (CLR) of multiple oral doses
Part 2: Physical Exams | Baseline up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in physical examinations
Part 2: ECGs | Baseline up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in ECGs
Part 2: Safety Labs | Baseline up to 14 days
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in safety labs
Part 2: Vitals Signs | Baseline up to 14 days
  Measure by number of subjects who experience potential clinically significant changes in vital signs
Part 3 CF: Physical Exams | Baseline up to 28 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in physical examinations
Part 3 CF: ECGs | Baseline up to 28 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in ECGs
Part 3 CF: Safety Labs | Baseline up to 28 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in safety labs
Part 3 CF: Vital Signs | Baseline up to 28 days
  Measured by number of subjects who experience potential clinically significant changes in vital signs
Part 4 CF: Physical Exams | Baseline up to 42 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in physical examinations
Part 4 CF: ECGs | Baseline up to 42 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in ECGs
Part 4 CF: Safety Labs | Baseline up to 42 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in safety labs
Part 4 CF: Vital Signs | Baseline up to 42 days
  Safety and tolerability measured by number of subjects who experience potential clinically significant changes in physical examinations

SECONDARY OUTCOMES:
Part 2: Apparent terminal half life (t1/2) of multiple oral doses PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 10
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in healthy adults
Part 2: Maximum plasma concentration (Cmax) of multiple oral doses PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 10
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in healthy adults
Part 2: Time to reach maximum plasma concentration (Tmax) of multiple oral doses PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 10
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in healthy adults
Part 2: AUC0-last of multiple oral doses when PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 10
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in healthy adults
Part 2: AUC from time 0 to infinity (AUC0-inf) of multiple oral doses when PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 10
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in healthy adults
Part 3 CF: Time to reach maximum plasma concentration (Tmax) of multiple oral doses PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 22
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in adults with CF
Part 3 CF: Maximum plasma concentration (Cmax) of multiple oral doses PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 22
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in adults with CF
Part 3 CF: AUC0-last of multiple oral doses when PTI 808 is co administered with PTI 801 and PTI 428 | Day 1 through Day 22
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 is co administered with PTI 801 and PTI 428 in adults with CF
Part 3 CF: FEV1 | Baseline through Day 28
  Change in forced expiratory volume in one second (FEV1) over time
Part 4 CF: Time to reach maximum plasma concentration (Tmax) of multiple oral doses of PTI 808 + PTI 801 co-administered with or without PTI 428 | Day 1 through Day 28
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 + PTI 801 is co administered with or with out PTI 428 in adults with CF
Part 4 CF: Maximum plasma concentration (Cmax) of multiple oral doses of PTI 808 + PTI 801 co-administered with or without PTI 428 | Day 1 through 28
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 + PTI 801 is co administered with or with out PTI 428 in adults with CF
Part 4 CF: AUC0-last of multiple oral doses when PTI 808 + PTI 801 is coadministered with or without PTI 428 in adults with CF | Day 1 through 28
  Evaluate the PK profile of PTI 808, PTI 801, and PTI 428 when PTI 808 + PTI 801 is co administered with or without PTI 428 in adults with CF
Part 4 CF: FEV1 | Baseline through Day 42
  Change in forced expiratory volume in one second (FEV1) over time
Part 4 CF Sweat Chloride | Baseline through Day 42
  Change in sweat chloride concentrations over time

OTHER OUTCOMES:
Part 2 Nasal biomarker | Baseline up to 14 days
  change in nasal epithelial mRNA and protein over time
Part 3 CF Sweat Chloride | Baseline up to 28 days
  Change in sweat chloride concentrations over time
Part 3 CF Nasal biomarker | Baseline up to 28 days
  Change in nasal epithelial mRNA and protein expression over time
Part 4 CF Weight and BMI | Baseline up to 42 days
  Change in weight and BMI over time
Part 4 CF Blood Glucose | Baseline up to 42 days
  Change in blood glucose over time
Part 4 CF disease-specific health related quality of life | Baseline up to 42 days
  Change in disease-specific health related quality of life over time
Part 4 CF Nasal biomarker | Baseline up to 42 days
  Change in nasal epithelial mRNA and protein expression over time

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Key, MD, Principal Investigator — ICON Early Phase Services (Parts 1 & 2); Patrick Flume, MD, Principal Investigator — Medical University of South Carolina (Parts 3 & 4)
Locations (48):
- United States (22):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine, University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Medical College, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - ICON Early Phase Services, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- John Hunter Hospital, Lambton, New South Wales, Australia
- Belgium (2):
  - Universitair ziekenhuis Brussel, Brussels
  - UZ Leuven, Leuven
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Québec
- University of Copenhagen Rigshospitalet, Copenhagen, Denmark
- France (6):
  - Hôpital Pasteur, Nice, Alpes-Maritimes
  - Hôpital Haut Lévêque, Pessac, Gironde
  - Hôpital Guillaume-et-René-Laennec, Nantes, Loire-Atlantique
  - Hôpital Maison Blanche Maladies respiratoires et allergologie, Reims, Marne
  - Hospices Civils de Lyon, Lyon
  - Hôpital Cochin, Paris
- Germany (5):
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Cologne, Cologne
  - Universitätsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universität, Frankfurt
  - Klinikum des Universität München, München
- Auckland Clinical Studies Ltd., Grafton, Auckland, New Zealand
- United Kingdom (6):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Western General Hospital, Edinburgh, Scotland
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Belfast City Hospital, Belfast
  - King's College Hospital, London
  - University Hospital Southampton, Southampton